CLINICAL TRIAL: NCT02404597
Title: Non-invasive Cardiac Output Monitoring in Patients With Burn Injuries
Brief Title: Cardiac Output Monitoring in Burn Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Potential participants have not yet been identified.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rachael Williams, Associate, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00078576
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Burns
Keywords: Cardiac output; Low blood pressure; Total Body Surface Area (TBSA)
MeSH Terms: conditions — Burns; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- NICOM (Experimental): Subjects with burns greater than 20% total body surface area (TBSA) will have a NICOM placed on them after the first 24 hours of admission if subject has an episode of hypotension (mean arterial pressure < 65 or a systolic blood pressure < 90mmHg). The NICOM will generate a number that reflects stroke volume of the heart. If the number is greater than 10 percent, subject will be given a bolus of crystalloid fluids. If the number is less than 10 percent, subject will start a medication to raise the blood pressure.
  Physicians may also use traditional endpoints of resuscitation include base deficit values and urine output goals of 0.5cc/kg/hr as indications of adequate intravenous fluid resuscitation.
  Interventions: Device: NICOM (non-invasive cardiac output monitor)
- Control (No Intervention): This is a retrospective comparison control group of patients with burns greater than 20% total body surface area (TBSA) admitted to the hospital from 7/1/2014-12/31/2014.

INTERVENTIONS:
Device: NICOM (non-invasive cardiac output monitor) — The non-invasive cardiac output monitor (NICOM) will be used to tailor fluid management to optimize resuscitation if the patient has an episode of hypotension (defined as systolic blood pressure <100 or mean arterial pressure <65). NICOM consists of two electrodes placed on the patient's chest and back and uses bioreactance technology to transduce signals to compute hemodynamic parameters on an associated monitor.
  The electrodes will remain on the patient for twenty minutes. Once the electrodes are in place the patient's leg will be raised to 45 degrees and the monitor to which the electrodes are attached will generate a number that reflects stroke volume of the heart. The electrodes will be removed once this number is determined.
  Arms: NICOM

SUMMARY:
The purpose of this study is to describe the use of non-invasive cardiac output monitors (NICOM) in patients with burn injuries and to develop a protocol for NICOM in a burn unit.

DETAILED DESCRIPTION:
Appropriate fluid resuscitation in the first 24 hours after a burn injury directly influences patient outcome and morbidity. Currently, there is some controversy surrounding the over and under-resuscitation and endpoints of resuscitation using older fluid resuscitation formulas in patients with burn injury. The NICOM has been used in the resuscitation of patients with sepsis. The NICOM will be used in patients with burn injury to determine the patient's fluid responsiveness and the need for additional fluid boluses versus medications to increase the patient's blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1) Burn greater than 20% TBSA (total body surface area)

Exclusion Criteria:

1) Burn less than 20% TBSA (total body surface area)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Total volume of fluid given | 24 hours
  The total volume of fluid given to the subjects in the first 24 hours
Rate of pressor use | Duration of hospital stay, an expected average of 30 days
  Defined as number of subjects that required pressor support (administration of cardiovascular supportive agents)

SECONDARY OUTCOMES:
Rate of pulmonary edema | Duration of hospital stay, an expected average of 30 days
  Defined as number of subjects with pulmonary edema
Rate of acute renal failure | Duration of hospital stay, an expected average of 30 days
  Defined as number of subjects with renal failure
Length of stay in intensive care unit (ICU) | 3 months
  Defined as the number of days from date of admission to date of first ICU discharge.
Length of hospital stay | 3 months
  Defined as the number of days from date of admission to date of first hospital discharge, regardless of if subject was discharged to home or other location.

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Williams, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States